CLINICAL TRIAL: NCT07302698
Title: Evaluation of the Pharmacokinetics and Onset Performance of Hezkue® Oral Sildenafil Suspension Following Alcohol Consumption in Healthy Adults
Brief Title: PK and Onset of Hezkue Oral Sildenafil Suspension After Alcohol Consumption
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aspargo Labs, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ASP-021-Sil
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-Arm Crossover (Experimental)
  Interventions: Drug: Hezkue Oral Sildenafil Suspension

INTERVENTIONS:
Drug: Hezkue Oral Sildenafil Suspension — Hezkue® oral sildenafil suspension will be administered as a single oral dose following controlled moderate alcohol consumption under fasting or standardized conditions, according to the study schedule, to evaluate pharmacokinetics, onset performance, and safety.

SUMMARY:
This is an open-label, randomized study evaluating the pharmacokinetics and onset performance of Hezkue® oral sildenafil suspension administered following moderate alcohol consumption in healthy adult subjects. Participants will receive Hezkue® under controlled alcohol-exposure conditions. Pharmacokinetic sampling, onset assessments, and safety evaluations will be conducted throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 21 to 55 years of age, inclusive.

Body mass index (BMI) between 18.0 and 30.0 kg/m², inclusive.

Medically healthy based on medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations, in the opinion of the investigator.

Able to safely consume moderate amounts of alcohol as judged by the investigator (for example, no history of alcohol intolerance, alcohol use disorder, or alcohol-related medical complications).

Blood pressure and heart rate within normal or non-clinically significant ranges at screening and baseline, in the opinion of the investigator.

Non-smoker or light smoker (10 cigarettes per day or fewer, or equivalent) willing to abstain during study confinement periods.

Able to understand and provide written informed consent before any study-specific procedures are performed.

Willing and able to comply with all study requirements, including alcohol restrictions, fasting, dosing schedules, and pharmacokinetic and onset assessments.

Females of childbearing potential must use acceptable contraception as determined by the investigator.

Exclusion Criteria:

* History or presence of any clinically significant cardiovascular disease, including but not limited to coronary artery disease, heart failure, clinically important arrhythmias, or uncontrolled hypertension or hypotension.

Resting systolic blood pressure or diastolic blood pressure, or heart rate, outside protocol-defined acceptable ranges at screening or baseline, in the opinion of the investigator.

Known hypersensitivity or contraindication to sildenafil, other phosphodiesterase type 5 (PDE5) inhibitors, alcohol, or any component of the study formulations.

Current or recent use of nitrates, nitric oxide donors, or guanylate cyclase stimulators (for example, riociguat).

History of significant hepatic, renal, gastrointestinal, neurologic, psychiatric, endocrine, hematologic, or respiratory disease that, in the investigator's opinion, could interfere with study participation or data interpretation.

History of syncope, significant orthostatic hypotension, or other conditions that may be worsened by sildenafil or alcohol.

History of alcohol use disorder, binge drinking patterns, or other substance use disorder, as determined by the investigator.

Positive urine drug screen or positive alcohol test at screening (outside scheduled alcohol administration for the study) or at admission.

Use of prescription or over-the-counter medications, herbal products, or dietary supplements within 14 days before the first study dose, unless considered acceptable by the investigator.

Positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV.

Participation in another clinical study or receipt of an investigational drug or device within 30 days or 5 half-lives (whichever is longer) before the first study dose.

Donation of 450 mL or more of blood, or significant blood loss, within 8 weeks before the first study dose.

Pregnant or breastfeeding females.

Women of childbearing potential not using acceptable contraception.

Any condition or circumstance that, in the opinion of the investigator, would make the participant unsuitable for the study or could interfere with compliance or study assessments.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve from Time Zero to Last Quantifiable Concentration (AUC₀-t) of Sildenafil | From predose up to approximately 24 hours postdose in each study period
Maximum Observed Plasma Concentration (Cmax) of Sildenafil | From predose up to approximately 24 hours postdose in each study period
Time to Onset of Effect as Assessed by Participant-Reported Onset | From dosing up to approximately 4 hours postdose in each study period

IPD SHARING:
Plan to Share IPD: No